CLINICAL TRIAL: NCT04685304
Title: Pharmacogenomics Applied to Chronic Pain Treatment in Primary Care
Acronym: PGx-ACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Kailos Genetics, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00002751
Record Dates: First submitted 2020-12-04; First posted 2020-12-28 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Chronic Pain
Keywords: pharmacogenetics; pharmacogenomics; CYP2D6; CYP2C9; tramadol; codeine; hydrocodone; NSAIDs; opioids
MeSH Terms: conditions — Chronic Pain | interventions — Pharmacogenomic Testing; Cytochrome P-450 CYP2D6; Cytochrome P-450 CYP2C9

STUDY DESIGN:
Intervention Model Description: An open-label, prospective, randomized trial design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGx-guided care (Experimental): Pharmacogenetic results (e.g., CYP2D6, CYP2C9) and a pharmacist consultation will be provided to their primary care provider. This consultation note (PharmD consult) will aid primary care providers in the interpretation and application of PGx results in prescribing decisions. The ultimate prescribing decision is at the discretion of the primary care provider and patient.
  Interventions: Genetic: Pharmacogenetic Testing; Other: Pharmacist Consultation Note
- Standard care (Active Comparator): Care for study subjects will occur without PGx results at the discretion of the study subject, their primary care provider.
  After the active participation ends (i.e. after the three month follow up is complete), PGx results and a PharmD consult will be provided similar to the PGx-guided arm.
  Interventions: Other: Delayed pharmacogenetic testing

INTERVENTIONS:
Genetic: Pharmacogenetic Testing — Genetic results will be reported for CYP2D6, CYP2C19, CYP2C9, CYP2B6, CYP3A4, CYP3A5, SLCO1B1, TPMT, and VKORC1.
  Other Names: pharmacogenomics; CYP2D6; CYP2C9; PGx
  Arms: PGx-guided care
Other: Pharmacist Consultation Note — Recommendations will be based on phenotypes translated from genetic data in accordance with CPIC guidelines. Drug interactions will be incorporated into phenotype assignments when appropriate.
  Arms: PGx-guided care
Other: Delayed pharmacogenetic testing — Pharmacogenetic testing and a pharmacist consultation note will be provided to participants provided to the standard care arm once 3 months have passed since their baseline visit.
  Arms: Standard care

SUMMARY:
Pharmacogenomics (PGx) Applied to Chronic pain Treatment in primary care (PGx-ACT) is an open-label, prospective, randomized trial. Participants prescribed a relevant opioid and meet additional eligibility criteria will be randomized into either a PGx-guided care (intervention) arm or standard care (control) arm. The investigators will test the hypothesis that patients with intermediate or poor CYP2D6 metabolism assigned to PGx-guided care arm will experience improved pain control at 3 months compared to patients in the standard care arm. Additionally, the study investigators will be evaluating non-pain related uses of PGx information in the chronic pain population.

DETAILED DESCRIPTION:
Chronic pain affects millions of Americans on an annual basis. Pharmacologic pain management strategies, which includes opioid analgesics, are widely used to treat chronic pain. The selection of an analagesic can be guided by pharmacogenomic (PGx) data via existing Clinical Pharmacogenetics Implementation Consortium (CPIC) guidelines. The rationale for PGx-guided treatment is based upon the CYP2D6 bioactivation of tramadol, codeine, and hydrocodone, whereas patients with reduced CYP2D6 function may not activate these drugs and therefore may not experience the effective treatment from these drugs. A prior pragmatic proof-of-concept trial testing the effects of CYP2D6-guided opioid prescribing on pain control provides additional evidence for this study.

This study is designed to evaluate the impact of PGx-guided treatment on chronic pain score improvement compared to standard conventional treatment in a pragmatic setting. It will test for multiple genes to enable incorporation of CPIC guidelines for other drugs (e.g., antidepressants, nonsteroidal antiinflammatory drugs), account for drug-drug interactions, and utilize recently updated CYP2D6 phenotype translation thresholds.

Primary objective: Identify the effects of providing pharmacogenomic (PGx) results and recommendations for patients with chronic pain who are treated in primary care clinics versus standard care.

Secondary objective: Explore non-pain related uses of PGx information in a population with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Any sex, 18 years of age or older
* Report chronic pain (i.e., pain for at least 3 months),
* Have a current prescription (prior to the enrollment visit) for either hydrocodone, tramadol, or codeine.
* This opioid is ordered by a provider associated with MedStar Health
* Treated at a participating primary care clinic (section 6)
* Willing and able to comply with scheduled visits, buccal sample collection, and other trial-related procedures.

Exclusion Criteria:

* Patients who have received a liver or bone marrow transplant.
* Patients with documented opioid use disorder (e.g., opioid use disorder on the problem list) or have current prescriptions for buprenorphine represent a level of complexity that are beyond the scope of this trial.
* Any surgical procedure that typically necessitates post-operative opioid (e.g., laparoscopic cholecystectomy, unilateral open and laparoscopic inguinal hernia repair, partial mastectomy with and without sentinel lymph node biopsy, uncomplicated cesarean delivery, minimally invasive hysterectomy, robotic retropubic prostatectomy, arthroscopic partial meniscectomy, and thyroidectomy) within the past 3 months or in the study period.
* Surgeries or procedures that would not typically require postoperative opioids are permissible (e.g., (uncomplicated vaginal delivery, cochlear implant, and cardiac catheterization).
* A urine drug screen at enrollment or during the study identifies the patient ingesting a narcotic medication that is not prescribed to them. It is not a study requirement that any patients have completed a urine drug screen as this will be considered part of clinical practice per the treating provider.
* Known to have previously received CYP2D6 testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2024-04-11 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity | 3 months
  The change in composite pain intensity among CYP2D6 poor or intermediate metabolizers between the baseline visit and 3 months. The composite pain intensity is defined as the mean of current, worst, and average pain intensity. The PROMIS Scale v1.0 Pain Intensity 3a will be used to collected pain intensity data. The scale asks three separate questions regarding how intense the patient's pain is on average over the past 7 days, at it's worst over the past 7 days, and at that moment. Options range from 1 (had no pain) to 5 (very severe).

SECONDARY OUTCOMES:
Opioid Use | 3 months
  The change number of morphine milliequivalents (MMEs) prescribed between baseline and 3 months.
Recommendation Acceptance | first encounter (baseline visit), 3 months, 12 months
  Proportion of patients with prescribing decisions concordant with PGx with recommendations
Significant Change in Pain Intensity | 3 months
  The proportion of patients with at least a 30% improvement in composite pain intensity.
Change in Physical Function | 3 months
  Using the PROMIS-29 Profile v2.0, assess the change in physical function between baseline and 3 months. The scale includes options that range from 1 (without any difficulty) to 5 (unable to do).
Change in Pain Interference Symptoms | 3 months
  Using the PROMIS-29 Profile v2.0, assess the change in symptoms between baseline and 3 months. The scale includes options that range from 1 (not at all) to 5 (very much).
Change in Pain Intensity Among Those with Therapy Concordant with PGx Recommendations | 3 months
  The subset of patients with actionable results (e.g., CYP2D6 poor or intermediate metabolism) will have pain intensity compared between those with therapy concordant and discordant with recommendations.
  The change in composite pain intensity between the baseline visit and 3 months. The composite pain intensity is defined as the mean of current, worst, and average pain intensity. The PROMIS Scale v1.0 Pain Intensity 3a will be used to collected pain intensity data. The scale asks three separate questions regarding how intense the patient's pain is on average over the past 7 days, at it's worst over the past 7 days, and at that moment. Options range from 1 (had no pain) to 5 (very severe).

CONTACTS AND LOCATIONS:
Overall Officials: Max Smith, PharmD, Principal Investigator — MedStar Health
Locations (1):
- MedStar Good Samaritan Hospital, Baltimore, Maryland, United States